CLINICAL TRIAL: NCT00715806
Title: Reduction of Claustrophobia During Magnetic Resonance Imaging: Randomized, Controlled Trial
Brief Title: Claustrophobia and Magnetic Resonance Imaging
Acronym: CLAUSTRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Marc Dewey, Charité
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: EA1/020/08
Record Dates: First submitted 2008-07-10; First posted 2008-07-15 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2009-11

CONDITIONS: Claustrophobia
Keywords: claustrophobia; magnetic resonance imaging; MRI; anxiety; open design; severely anxious patients
MeSH Terms: conditions — Claustrophobia; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Device: Open MRI scanner.
- 2 (Active Comparator)
  Interventions: Device: Closed MRI scanner.

INTERVENTIONS:
Device: Open MRI scanner. — Imaging in an Open MRI scanner.
  Arms: 1
Device: Closed MRI scanner. — Imaging in a short-bore closed MRI scanner.
  Arms: 2

SUMMARY:
The objective of the study is to determine the ability of open magnetic resonance imaging (MRI) scanners to reduce claustrophobic reactions, thereby enabling more examinations of severely anxious patients. The investigators hypothesize that anxiety-based claustrophobia that prevents MR examinations without sedation can be reduced using an open MR scanner design thereby improving clinical management of those patients.

ELIGIBILITY:
Inclusion Criteria:

* Severely anxious patients with reported claustrophobia during MRI or with the inability to undergo MR examinations on conventional scanners
* Clinical indication for MR imaging of the head, spine, or shoulder.

Exclusion Criteria:

* Contraindication to MR imaging (shrapnells, pacemakers, certain unsafe implants)
* Age below 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
The ability of an open MRI scanner to reduce claustrophobic reactions that prevent MR examinations. | Before or During MRI

SECONDARY OUTCOMES:
Impact of MR imaging results on subsequent measurement. | 6 months after MRI

CONTACTS AND LOCATIONS:
Overall Officials: Marc Dewey, MD, Principal Investigator — Charité
Locations (1):
- Charité, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] Dewey M, Schink T, Dewey CF. Claustrophobia during magnetic resonance imaging: cohort study in over 55,000 patients. J Magn Reson Imaging. 2007 Nov;26(5):1322-7. doi: 10.1002/jmri.21147. PMID 17969166
- [Background] Dewey M, Schink T, Dewey CF. Frequency of referral of patients with safety-related contraindications to magnetic resonance imaging. Eur J Radiol. 2007 Jul;63(1):124-7. doi: 10.1016/j.ejrad.2007.01.025. Epub 2007 Mar 23. PMID 17383136
- [Background] Enders J, Zimmermann E, Rief M, Martus P, Klingebiel R, Asbach P, Klessen C, Diederichs G, Bengner T, Teichgraber U, Hamm B, Dewey M. Reduction of claustrophobia during magnetic resonance imaging: methods and design of the "CLAUSTRO" randomized controlled trial. BMC Med Imaging. 2011 Feb 10;11:4. doi: 10.1186/1471-2342-11-4. PMID 21310075
- [Derived] Enders J, Rief M, Zimmermann E, Asbach P, Diederichs G, Wetz C, Siebert E, Wagner M, Hamm B, Dewey M. High-field open versus short-bore magnetic resonance imaging of the spine: a randomized controlled comparison of image quality. PLoS One. 2013 Dec 31;8(12):e83427. doi: 10.1371/journal.pone.0083427. eCollection 2013. PMID 24391767
- [Derived] Enders J, Zimmermann E, Rief M, Martus P, Klingebiel R, Asbach P, Klessen C, Diederichs G, Wagner M, Teichgraber U, Bengner T, Hamm B, Dewey M. Reduction of claustrophobia with short-bore versus open magnetic resonance imaging: a randomized controlled trial. PLoS One. 2011;6(8):e23494. doi: 10.1371/journal.pone.0023494. Epub 2011 Aug 22. PMID 21887259